CLINICAL TRIAL: NCT02799927
Title: A Split-mouth Trial Comparing Biodentine and Calcium Hydroxide in the Indirect Pulp Treatment on Primary Teeth
Brief Title: Comparison Between Biodentine and Calcium Hydroxide in the Indirect Pulp Treatment on Primary Teeth
Acronym: IPT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: José Arturo Garrocho Rangel (Other)
Responsible Party: Sponsor-Investigator, José Arturo Garrocho Rangel, Professor/Lecturer, Universidad Autonoma de San Luis Potosí
Organization: Universidad Autonoma de San Luis Potosí (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEI-FE-003-014
Record Dates: First submitted 2016-05-19; First posted 2016-06-15 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Dental Caries
Keywords: Indirect Pulp Treatment; Primary Teeth; Biodentine; Calcium Hydroxide; Split-Mouth design
MeSH Terms: conditions — Dental Caries | interventions — tricalcium silicate; Calcium Hydroxide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biodentine (Experimental): Biodentine (Septodont, Saint-Maur-des-Fosses, France) has been recently introduced and marketed as a bioactive dentin substitute. The Biodentine powder contains tricalcium silicate, dicalcium silicate and calcium oxide, while its liquid consists of calcium chloride and a carboxylate-based hydrosoluble polymer (water-reducing agent).
  After local anesthesia and rubber dam isolation, carious peripheral dentin is eliminated with a high speed tungsten-carbide bur # 3, and air-water spray. Then, the cavity's floor soft dentin layer is carefully removed with a sharply-edged sterilized hand excavator, leaving only the hard dentin adjacent to the pulp ceiling. The cavity is thoroughly rinsed only with water and dried with sterilized cotton pellets. The next step consists in the preparation of Biodentine liner (a mix of powder and liquid), following the manufacturers' instructions, and its placement over the remanent carious dentin layer.
  Interventions: Procedure: Indirect Pulp Treatment with Bioactive Dentin Substitute
- Ultra-Blend plus (Calcium hydroxide) (Active Comparator): Ultra-Blend plus® (Ultradent Products Inc., South Jordan, UT, USA). This material is a light-activated calcium hydroxide based-liner. Calcium hydroxide has demonstrated to reduce and promote immediate deactivation of the residual microorganisms after IPT.
  After local anesthesia and rubber dam isolation, carious peripheral dentin is eliminated with a high speed tungsten-carbide bur # 3, and air-water spray. Then, the cavity's floor soft dentin layer is carefully removed with a sharply-edged sterilized hand excavator, leaving only the hard dentin adjacent to the pulp ceiling. The cavity is thoroughly rinsed only with water and dried with sterilized cotton pellets. The next step consists in the placement of Ultra-Blend plus liner over the remanent carious dentin layer, using a dycal metallic applicator. Finally, the liner is cured through light exposure during 20 seconds .
  Interventions: Procedure: Indirect Pulp treatment with Calcium hydroxide

INTERVENTIONS:
Procedure: Indirect Pulp Treatment with Bioactive Dentin Substitute — The indirect pulp treatment (IPT), with Biodentine is a vital pulp procedure for dep cariously primary teeth without carious exposure, involving the removal of the softened, humid and infected dentin layer, leaving intact intentionally the deepest layer of the dentin-pulp complex, followed by the placement of Biodentine and a hermetic restoration to provide a seal against microleakage, without the necessity to reenter for removing the residual caries.
  Other Names: Biodentine
  Arms: Biodentine
Procedure: Indirect Pulp treatment with Calcium hydroxide — The indirect pulp treatment (IPT), with Biodentine is a vital pulp procedure for dep cariously primary teeth without carious exposure, involving the removal of the softened, humid and infected dentin layer, leaving intact intentionally the deepest layer of the dentin-pulp complex, followed by the placement of Ultra-Blend plus, and a hermetic restoration to provide a seal against microleakage, without the necessity to reenter for removing the residual caries.
  Other Names: Ultra-Blend plus
  Arms: Ultra-Blend plus (Calcium hydroxide)

SUMMARY:
Objective: The study's main purpose is to evaluate and compare the clinical and radiographic outcomes of Biodentine and a light-activated calcium hydroxide based-liner (Ultra-Blend plus®) as indirect pulp treatment (IPT) liners, over the dentin-pulp complex of vital primary molars with carious lesions approaching the pulp. Study design: 80 four-to-eight year-old patients were enrolled from a Mexican University Pediatric Dentistry Clinic. A split-mouth design trial is being conducted in order to compare both IPT interventions on 160 bilateral primary teeth, without signs or symptoms of irreversibly inflamed or degenerative pulp tissue. Teeth were treated and restored with a preformed crown in a single session, and then closely followed-up for 1, 3, 6, 12, 18, and 24 months.

DETAILED DESCRIPTION:
A Split-mouth clinical trial was the design selected. Clinical Procedures: IPT procedures were carried out by three pediatric dentistry residents (E.K.C.G., R.A.V.V., and J.M.A.R.), previously trained in the clinical setting with a pilot sample of 10 similar child patients each. Study participants received local anesthesia and rubber dam isolation, which was disinfected, followed by the remove of the carious peripheral dentin with high speed tungsten-carbide bur # 3, and air-water spray. Then, the soft dentin layer was carefully removed with a sharply-edged sterilized hand excavator, based on tactile and visual standards, leaving only the hard dentin adjacent to the pulp ceiling. The cavity was thoroughly rinsed only with water and then dried with sterilized cotton pellets; no other special disinfection protocol was applied. The next step consisted in the placement of the correspondent liner over the remanent carious dentin layer, following the manufacturers' instructions, and according to the randomly assignment scheme previously described. In the case of the control group, the liner was cured undr 20 seconds of light exposure. All treated molar were restored with stainless steel preformed crowns (3M ESPE) cemented with glass ionomer (Ketac-Cem, 3M ESPE). One week later, the same procedure was repeated in the opposite tooth with the contrary IPT agent.

ELIGIBILITY:
Inclusion criteria:

* At least one restorable first or second primary molar in each side of the mouth, affected by an occlusal cavitated active caries lesion in deep dentin.
* Cooperative patients.
* Participants were included in the trial after parental acceptance through a signed informed consent.

Exclusion criteria:

* Molars with mobility, spontaneous pain or fistula, and radiographic findings such as a carious lesion with no evidence of residual dentin over the pulp chamber or manifest pulp exposition.
* Normally internal root resorption or physiological root resorption less than 1/3.
* Presence of periradicular/furcal radiolucent lesions.
* Occurrence of a carious pulp exposure and bleeding during the operative procedure.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-04 (Actual); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Pain. Binary variable (present/absent). | 2 years
  Pain is assessed through interrogatory. It is a binary variable (pain present or pain absent)

SECONDARY OUTCOMES:
Sensitivity to percussion. Binary variable (present/absent). | 2 years
  Treated tooth is softly hit with a dental handle mirror. Sensitivity is recorded as a binary variable (present/absent).
Abnormal tooth mobility. Binary variable (present/absent). | 2 years
  This variable is measured by handling the treated tooth with two fingers. It is a binary variable (present/absent).
Soft tissues inflammation. Binary variable (present/absent). | 2 years
  This feature is assessed through visual examination of surrounding soft gingival tissues (texture, color, size). It is a binary variable(present/absent) .
Periradicular lesions. Binary variable (present/absent). | 2 years
  These lesions are observed through radiographic examination. They appear as radiolucencies around the tooth's root (s). It is a binary variable (present/absent)
Sensitivity to palpation. Binary variable (present/absent). | 2 years
  Treated tooth is softly pressed with a finger. Sensitivity is recorded as a binary variable (present/absent).

CONTACTS AND LOCATIONS:
Overall Officials: María S Ruiz, M. Sc., Study Chair — Pediatric Dentistry Postgraduate Program

IPD SHARING:
Plan to Share IPD: Undecided
Yes. Only in case of future systematic reviews with meta-analysis.

REFERENCES:
- [Background] Al-Zayer MA, Straffon LH, Feigal RJ, Welch KB. Indirect pulp treatment of primary posterior teeth: a retrospective study. Pediatr Dent. 2003 Jan-Feb;25(1):29-36. PMID 12627699
- [Background] Casagrande L, Bento LW, Rerin SO, Lucas Ede R, Dalpian DM, de Araujo FB. In vivo outcomes of indirect pulp treatment using a self-etching primer versus calcium hydroxide over the demineralized dentin in primary molars. J Clin Pediatr Dent. 2008 Winter;33(2):131-5. doi: 10.17796/jcpd.33.2.82r1tp71x75m5345. PMID 19358380
- [Background] Fernandes JM, Massoni AC, Ferreira JM, Menezes VA. Use of calcium hydroxide in deep cavities of primary teeth. Quintessence Int. 2013;44(6):417-23. doi: 10.3290/j.qi.a29503. PMID 23534045
- [Background] Kim J, Song YS, Min KS, Kim SH, Koh JT, Lee BN, Chang HS, Hwang IN, Oh WM, Hwang YC. Evaluation of reparative dentin formation of ProRoot MTA, Biodentine and BioAggregate using micro-CT and immunohistochemistry. Restor Dent Endod. 2016 Feb;41(1):29-36. doi: 10.5395/rde.2016.41.1.29. Epub 2016 Jan 4. PMID 26877988
- [Background] Petrou MA, Alhamoui FA, Welk A, Altarabulsi MB, Alkilzy M, H Splieth C. A randomized clinical trial on the use of medical Portland cement, MTA and calcium hydroxide in indirect pulp treatment. Clin Oral Investig. 2014;18(5):1383-9. doi: 10.1007/s00784-013-1107-z. Epub 2013 Sep 17. PMID 24043482
- [Background] Trairatvorakul C, Sastararuji T. Indirect pulp treatment vs antibiotic sterilization of deep caries in mandibular primary molars. Int J Paediatr Dent. 2014 Jan;24(1):23-31. doi: 10.1111/ipd.12022. Epub 2013 Jan 24. PMID 23346907